CLINICAL TRIAL: NCT02600273
Title: Novel Approaches to Reducing Tobacco Related Harm Among HIV-Infected Smokers
Brief Title: Novel Approaches to Reducing Tobacco Related Harm
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: Pro00067757; 5P30AI064518 (NIH)
Record Dates: First submitted 2015-11-05; First posted 2015-11-09 (Estimated); Last update posted 2020-09-30 (Actual); Status verified 2020-09

CONDITIONS: Smoking; Tobacco Smoking Behavior; Cigarette Smoking
MeSH Terms: conditions — Smoking; Cigarette Smoking

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Usual brand cigarettes (Active Comparator): During one session, participants will smoke their usual brand cigarettes
  Interventions: Other: Usual brand cigarettes
- Lower nicotine content cigarettes (Experimental): During one session, participants will smoke SPECTRUM Research Cigarettes
  Interventions: Other: Lower nicotine content cigarettes
- Electronic cigarettes 1 (Experimental): During one session, participants will use an electronic cigarette with 0 mg/mL nicotine e-liquid
  Interventions: Other: Electronic cigarettes 1
- Electronic cigarettes 2 (Experimental): During one session, participants will use an electronic cigarette with 18 mg/mL nicotine e-liquid
  Interventions: Other: Electronic cigarettes 2

INTERVENTIONS:
Other: Usual brand cigarettes — Usual brand cigarettes
  Arms: Usual brand cigarettes
Other: Lower nicotine content cigarettes — SPECTRUM research cigarettes
  Arms: Lower nicotine content cigarettes
Other: Electronic cigarettes 1 — Electronic cigarette with 0 g/mL e-liquid
  Arms: Electronic cigarettes 1
Other: Electronic cigarettes 2 — Electronic cigarette with 18 g/mL e-liquid
  Arms: Electronic cigarettes 2

SUMMARY:
The purpose of this study is to assess initial reactions to alternative nicotine/tobacco products among smokers living with HIV.

DETAILED DESCRIPTION:
Participants will sample 4 alternative nicotine/tobacco products and provide initial reactions to the products.

ELIGIBILITY:
Inclusion Criteria:

1. HIV-infected adults age 18 and older currently receiving HIV care
2. Self-report smoking ≥10 cigarettes/day of a brand delivering >0.5mg nicotine for >2yrs
3. Have afternoon expired CO concentrations of ≥10ppm or morning urinary cotinine >100ng/ml (as measured with NicAlert)

Exclusion Criteria:

1. Impaired mental status as assessed by observation
2. Acute intoxication as measured by breath alcohol level (BAL) > 0
3. Current use of nicotine replacement or other pharmacotherapy for smoking cessation
4. Previous use of e-cigarettes
5. Use of other tobacco products (e.g., chew tobacco, cigars) on > 10 of the past 30 days
6. Unstable HIV or associated comorbidities, as determined by a licensed medical professional.
7. Pregnancy (Females testing positive for pregnancy and any participants wishing to quit immediately will be referred to community smoking cessation treatment and will be excluded from the study)
8. Blood pressure at or above 160/100 or below 90/50
9. Heart rate at or above 105 bpm or below 45 bpm

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2019-06 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
Subjective effects, as measured by survey | within 2 minutes after sampling product(s)
  Satisfaction, acceptability, withdrawal, craving
Risk perceptions, as measured by survey | Before and within 2 minutes after sampling product(s)
  Risk perceptions of products
Interest and confidence in quitting, as measured by survey | within 2 minutes after sampling product(s)
  Interest and confidence in using and purchasing the tested products in the future

SECONDARY OUTCOMES:
Reinforcing properties of product(s), as measured by survey | within 2 minutes after sampling product(s)
  Behavioral economics measures (commodity purchase task & cross-price elasticity)

CONTACTS AND LOCATIONS:
Overall Officials: F. Joseph McClernon, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University School of Medicine, Durham, North Carolina, United States